CLINICAL TRIAL: NCT05481268
Title: Comparative Efficacy of Kinesiotaping and Stretching on Sternocleidomastoid and Upper Trapezius Muscles in Patients Suffering From Myofascial Pain Due to Temporomandibular Joint Disorder
Brief Title: Kinesiotaping and Stretching on SKM and Upper Trapezius Muscle in TMD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Ozge Baykan Copuroglu, Prelector/ Physiotherapist, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulArelUTME
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: TMJ Disc Disorder; Myofascial Pain
Keywords: Temporomandibular pain; Kinesiotape; Stretching
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiotaping Group (Experimental): In the Kinesiotaping Group patients had muscle technique-inhibition method. An 'I' shaped tape was used for both SCM and upper trapezius.
  Interventions: Other: Kinesiotaping Group
- Stretching Group (Experimental): The patient was stretched in a relaxed and supported position and physiotherapist positioned the patient passively for stretching.
  Interventions: Other: Stretching Group
- Control Group (Other): Control Group patients, after the assessment by the dentist, the treatment method approved by the dentist was performed.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Kinesiotaping Group — In the Kinesiotaping Group patients had muscle technique-inhibition method. An 'I' shaped tape was used for both SCM and upper trapezius. The tension of the tape was adjusted between 20 and 25% and the application was performed in the longest position of the muscle. The inhibition technique was applied from the insertion to the origin of the muscle. The tape was applied to cover the trigger points where pain was felt. For upper trapezius, the muscle was taped in the opposite direction on the cervical region in lateral flexion, slight flexion, shoulder depression and using the muscle technique with the I tape. For SCM muscle, the tape was applied on the muscle in the opposite direction on the cervical region with positioning in lateral flexion, extension and ipsilateral rotation using the muscle technique with I tape Taping was applied every 3 days and totally in 4 cycles.
  Arms: Kinesiotaping Group
Other: Stretching Group — In our application, 3 cycles of 20 seconds of stretches were applied to upper trapezius and SCM muscle. The patient was stretched in a relaxed and supported position and physiotherapist positioned the patient passively for stretching. For the SCM muscle, stretching was achieved in the positions of contralateral lateral flexion, ipsilateral rotation and extension. For upper trapezius, stretching was performed in flexion and lateral flexion. Stretching was performed every 3 days in 4 cycles in total.
  Arms: Stretching Group
Other: Control Group — Control Group patients, after the assessment by the dentist, the treatment method approved by the dentist was performed. The assessment was performed before treatment, at the end of week 1 and at the end of week 2.
  Arms: Control Group

SUMMARY:
Purpose: This study determined the effects of Kinesiotaping and Stretching on pain, cervical joint range of motion and functional status in patients with myofascial pain due to temporomandibular joint disorder.

Methods: 33 patients with myofascial pain due to temporomandibular joint disorder were included in the study. The patients were divided into three groups by simple randomization (Kinesiotaping group, Stretching group and Control group). Patients in the Kinesiotaping and Stretching groups received application for their Upper Trapezius and Sternocleidomastoid muscles twice a week for two weeks by the same physiotherapist. No application was made to the Control group. Cervical joint range of motion, muscle strength and pain were evaluated. Additionally, algometry tests and functional evaluation were performed. The tests were performed in the Kinesiotaping and Stretching groups before the applications and at the end of week 1 and week 2, on the other hand Control group evaluated before the application and at the end of week 2.

DETAILED DESCRIPTION:
This study is my master's thesis that I conducted in 2018. Our prospective clinical study was approved by the Non-Interventional Ethics Committee. The study was conducted at Dentistry Prosthetic Odontotherapy Outpatient Clinic between February 2018 and April 2018. Volunteering 33 patients between the ages of 18 to 60 years and who applied clinics and were diagnosed with myofascial pain due to TMJ disorder according to Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) classification were included in the study. The patients were divided into groups using simple randomization method. There are 11 patients in groups. Blinding was ensured by patients and dentist were unaware the type of physiotherapy treatment application. Patient evaluation was repeated 3 times: before the treatment, at the end of week 1, and at the end of week 2 of the treatment.

In our study, the effects of conservative treatment options used in 'treatment of TMD on 'disease symptoms were examined compared with the control group. A 2-week follow-up was foreseen for the acute impact outcomes of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Myofascial pain according to RDC/TMD
* Natural posterior occlusion and volunteering
* Being informed and signing the consent to participate in the research.

Exclusion Criteria:

* Presence of dentofacial anomalies
* Arthralgia
* Disk displacement
* General inflammatory connective tissue diseases (e.g. rheumatoid arthritis)
* Psychiatric disease
* Tumor
* Orofacial disease symptoms (neuralgia, migraine, etc.)
* Local skin infection
* Using regular analgesic
* Fibromyalgia
* History of TMJ-related surgery
* Findings of allergy related to Kinesiotape.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 2 weeks
  The subjective pain intensity of the patients was assessed with the Visual Analogue Scale. The Visual Analog Scale includes scoring between 0 and 10. The corresponding numbers from 0 to 10 were explained to the patients. It was explained that the absence of pain was 0, the most severe pain felt was 10, and moderate pain was 5. For the Upper Trapezius and SCM muscle, the patients were asked to mark their resting and functional pain from the scale.Additionally, pain during palpation of the upper trapezius and sternocleidomastoid muscle was assessed with algometry.
Range of Motion | 2 weeks
  The range of motion of the cervical joint was assessed using a goniometer
Research Diagnostic Criteria for Temporomandibular Disorders | 2 week
  Klinik değerlendirme formunun içeriğinde ağrının nedeni ve ağrının tarafı, ağız açılma şekli ve açılma miktarı, eklem sesleri, eksantrik hareket miktarları ve hareket sırasındaki ağrı durumları, eklem sesleri ve kas ağrıları palpasyonla değerlendirildi. .
Muscle Strength | 2 week
  Cervical muscle strength was assessed manually
Mouth Opening Distance | 2 weeks
  The mouth opening of the patients was measured in millimeters for the distance between anterior incisors of the upper and lower jaws.

SECONDARY OUTCOMES:
The Patient Health Questionnaire | 2 weeks
  The Patient Health Questionnaire was used for comparison in the assessments are two of the subtests of the RDC/TMD questionnaire. The purpose of those tests was to obtain numerical data and to observe the comparison objectively.
Jaw Functional Limitation Scale | 2 weeks
  It has three levels of functional limitation, including chewing (6 items), jaw mobility (4 items), and verbal and emotional expression (10 items). Each item is rated on a numeric rating scale from 0 to 10. 0, no limitation; 10 indicates severe limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Baykan Copuroglu, MSc, Principal Investigator — Istanbul Arel University
Locations (1):
- Arel University, Istanbul, Turkey (Türkiye)